CLINICAL TRIAL: NCT06449820
Title: Janus Kinase Inhibitors for the Treatment of Acute Severe Ulcerative Colitis: a Retrospective Cohort Study
Brief Title: Janus Kinase Inhibitors for the Treatment of Acute Severe Ulcerative Colitis
Acronym: ATTRACT
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Dr Laurent PEYRIN-BIROULET, Principal Investigator / Scientific responsible, Central Hospital, Nancy, France
Other Study IDs: 2024PI030
Record Dates: First submitted 2024-04-15; First posted 2024-06-10 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ulcerative colitis (UC) is an incurable, immune-mediated inflammatory disease of the large bowel that typically requires long term immunosuppressive drugs to induce and maintain remission. Hospitalisation due to severe, uncontrolled disease is a common occurrence and estimated to affect up to 25% of UC patients. Janus kinase inhibitors (JAKi) have attracted considerable attention as potential candidates for treating hospitalised patients with severe UC and are increasingly used in this setting. For tofacitinib, there are accumulating data supporting their use as effective induction agents to prevent colectomy and reduce length of hospitalisation, however, these are limited to small case series and small cohort studies only. There are no published data for the use of filgotinib and upadacitinib for treating severe inpatient colitis.

The aim of this study is to develop a large retrospective cohort of JAKi-treated hospitalised UC patients to describe the safety and effectiveness of using JAKi in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old,
* Established diagnosis of ulcerative colitis as per ECCO (European Crohn´s and Colitis Organisation) criteria,
* Hospitalisation at any point for treatment of ulcerative colitis disease relapse,
* Receiving at least one dose of tofacitinib, filgotinib, or upadacitinib for the treatment of severe UC during inpatient stay,
* Endoscopically confirmed active disease (Mayo endoscopic subscore ≥ 2) within previous four weeks,
* Patient who has received full information about the organization of the research and who has not objected to his or her participation and to the use of his or her data.

Exclusion Criteria:

* Diagnosis of Crohn's disease or unclassified Inflammatory Bowel Disease,
* Receiving JAKi prior to admission,
* Clostridium difficile, cytomegalovirus (CMV), or other enteric infections identified on admission.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for ulcerative colitis disease relapse and treated during their stay with JAKi (tofacitinib, filgotinib, or upadacitinib) between 01/01/2019 and 01/12/2023.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Treatment failure up to day 98 after JAKi initiation to describe treatment effectiveness | after study completion, average of 1 month
  * Absence of steroid-free clinical remission according to the PRO-2 (stool ≤1 and rectal bleeding sub-score of 0)
  * Use of a prohibited treatment for relapse (partial Mayo score >5)
  * Severe adverse event leading to discontinuation of JAKi treatment
  * Colectomy
  * Death during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy University Hospital, Vandœuvre-lès-Nancy, Sélectionnez Un Département / État, France

IPD SHARING:
Plan to Share IPD: Undecided